CLINICAL TRIAL: NCT02755376
Title: A Randomized, Single Center, Investigator Initiated Clinical Trial to Evaluate Enhancement of Healing Between Bone Tunnel and Graft in Anterior Cruciate Ligament (ACL) Injury Using Human Umbilical Cord Blood Derived Mesenchymal Stem Cell
Brief Title: Development of Novel Strategy for Treatment of Anterior Cruciate Ligament (ACL) Injury Using Stem Cell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC 2013-07-117-002
Record Dates: First submitted 2015-02-22; First posted 2016-04-28 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2018-12

CONDITIONS: Deficiency of Anterior Cruciate Ligament
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACL reconstruction only (Active Comparator): only ACL reconstruction without any injection
  Interventions: Procedure: ACL reconstruction only
- ACL reconstruction + Cartistem(TM) (Experimental): ACL reconstruction and concomitant Cartistem(TM) injection which is human cord blood derived mesenchymal stem cell under arthroscopy.
  Interventions: Biological: Cartistem(TM); Procedure: ACL reconstruction only
- ACL reconstruction + Hyaluronic acid (Experimental): ACL reconstruction and concomitant hyaluronic acid injection under arthroscopy
  Interventions: Biological: hyaluronic acid; Procedure: ACL reconstruction only

INTERVENTIONS:
Biological: Cartistem(TM) — ACL reconstruction and injection of Cartstem(TM), human cord blood derived mesenchymal stem cell under arthroscopy.
  Arms: ACL reconstruction + Cartistem(TM)
Biological: hyaluronic acid — ACL reconstruction and injection of hyaluronic acid under arthroscopy.
  Arms: ACL reconstruction + Hyaluronic acid
Procedure: ACL reconstruction only — ACL reconstruction only without any injection under arthroscopy

SUMMARY:
Purpose:Development of novel strategy for treatment of anterior cruciate ligament (ACL) injury using stem cell.

DETAILED DESCRIPTION:
1. Purpose: Development of novel strategy for treatment of anterior cruciate ligament (ACL) injury using stem cell.
2. Subject: Anterior cruciate ligament (ACL) injury 30 patients

   * ACL reconstruction: 10
   * ACL reconstruction + Human cord blood derived mesenchymal stem cells and hyaluronic acid (Cartistem (TM)): 10
   * ACL reconstruction + hyaluronic acid: 10
3. Hypothesis: Human Cord blood derived mesenchymal stem cells can enhance healing between bone tunnel and graft in ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20~50
2. Lachman test grade II,III or Pivot shift test grade I,II,III or ACL rupture in MRI
3. prothrombin time (PT) (INR) <1.5, activated partial thromboplastin time (aPTT) <1.5 x control
4. Creatinine ≤2.0 ㎎/㎗, protein uria(dipstick) ≤ trace
5. Bilirubin ≤2.0 ㎎/㎗, aspartate aminotransferase (AST) /Alanine Aminotransferase (ALT) ≤100 IU/L
6. No surgery and radiation therapy in recent 6 weeks
7. No pregnancy
8. No combine ligament instability ≥ grade II in physical examination (grade 0: none, grade I: 0~5mm, grade II: 5~10mm, grade III: >10mm)
9. voluntary singed a consent form

Exclusion Criteria:

1. Degenerative osteoarthritis in knee
2. Revision or other surgery history (stem cell treatment)
3. Chronic inflammatory joint disease like rheumatoid arthritis
4. Infectious disease need to administration of parenteral antibiotics
5. Autoimmune disease
6. Myocardial infarction, congestive heart failure, other serious heart disease
7. Uncontrolled hypertension
8. Serious medical disease
9. Pregnancy and breast-feeding
10. psychiatric disorder and epilepsy
11. Alcohol overuse
12. Smoking overuse
13. Administration of immunosuppressive agents like Cyclosporin A or Azathioprine in recent 6 weeks prior screening test
14. Patient participating in other clinical trials in recent 4 weeks
15. Combined ligament instability ≥ grade II in physical test.
16. No allergy history to gentamicin antibiotics
17. Hypersensitivity patient to bovine protein, hyaluronic acid, and anesthetic agent
18. Inappropriate patient judged by researcher.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Bone formation on interface between bone tunnel and graft | Changes at 12 week, 24 week, 48 week after surgery

SECONDARY OUTCOMES:
Arthroscopic grading of graft | 48 week after surgery
Telos stress X-ray | Changes at 12 week, 24 week, 48 week after surgery
KT-2000 | Changes at 12 week, 24 week, 48 week after surgery
clinical knee scoring | Changes at 12 week, 24 week, 48 week after surgery
Instability assessing with physical examination | Changes at 12 week, 24 week, 48 week after surgery
Tunnel enlargement after anterior cruciate ligament reconstruction | Changes at 12 week, 24 week, 48 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joon Ho Wang, MD, Ph D, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
age, physical exam, lab, etc will be shared